CLINICAL TRIAL: NCT06097754
Title: Intermittent Exogenous Ketosis (IEK): A Novel Strategy to Improve Hypoxic Tolerance and Adaptation
Brief Title: Intermittent Exogenous Ketosis (IEK) at High Altitude
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jozef Stefan Institute (Other)
Collaborators: KU Leuven (Other); University of Lausanne (Other)
Responsible Party: Principal Investigator, Tadej Debevec, Principal Investigator, Jozef Stefan Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IEK Weave
Record Dates: First submitted 2023-10-13; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Ketosis; Hypoxia
Keywords: Acclimatization; Altitude; Cardiorespiratory; Cerebrovascular; Exercise; Ketone; Acute Mountain Sickness; Sleep; Cognitive
MeSH Terms: conditions — Ketosis; Hypoxia; Motor Activity; Altitude Sickness | interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Intervention Model Description: 1 group with ketone ester supplementation and 1 group with taste and viscosity matched placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone group (Experimental): Ketone esters will be provided
  Interventions: Dietary Supplement: Ketone ester
- Control (Placebo Comparator): Ketone placebo will be provided
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone ester — Ketone ester: A total of 300g ketone ester supplementation will be provided in one of the 72h experimental sessions in order to establish intermittent exogenous ketosis. Sucralose (5% w/w) is added to the ketone ester (R)-3-hydroxybutyl (R)-3-hydroxybutyrate
  Hypobaric hypoxia: 72 hours experimental protocol conducted at terrestrial altitude
  Arms: Ketone group
Dietary Supplement: Placebo — Placebo: Water, 5% sucralose (w/w), octaacetate (1 mM)
  Hypobaric hypoxia: 72 hours experimental protocol conducted at terrestrial altitude
  Arms: Control

SUMMARY:
Altitude-related hypoxia decreases human functional capacity, especially during exercise. Even with prolonged acclimatization, the physiological adaptations are insufficient to preserve exercise capacity, especially at higher altitudes completely. Consequently, there has been an ongoing search for various interventions to mitigate the negative effects of hypoxia on human performance and functional capacity. Interestingly, early data in rodents and humans indicate that intermittent exogenous ketosis (IEK) by ketone ester intake improves hypoxic tolerance, i.e.by facilitating muscular and neuronal energy homeostasis and reducing oxidative stress. Furthermore, there is evidence to indicate that hypoxia elevates the contribution of ketone bodies to adenosine-triphosphate (ATP) generation, substituting glucose and becoming a priority fuel for the brain. Nevertheless, it is reasonable to postulate that ketone bodies might also facilitate long-term acclimation to hypoxia by upregulation of both hypoxia-inducible factor-1α and stimulation of erythropoietin production.

The present project aims to comprehensively investigate the effects of intermittent exogenous ketosis on physiological, cognitive, and functional responses to acute and sub-acute exposure to altitude/hypoxia during rest, exercise, and sleep in healthy adults. Specifically, we aim to elucidate 1) the effects of acute exogenous ketosis during submaximal and maximal intensity exercise in hypoxia, 2) the effects of exogenous ketosis on sleep architecture and quality in hypoxia, and 3) the effects of exogenous ketosis on hypoxic tolerance and sub-acute high-altitude adaptation. For this purpose, a placebo-controlled clinical trial (CT) in hypobaric hypoxia (real high altitude) corresponding to 3375 m a.s.l. (Rifugio Torino, Courmayeur, Italy) will be performed with healthy individuals to investigate both the functional effects of the tested interventions and elucidate the exact physiological, cellular, and molecular mechanisms involved in acute and chronic adaptation to hypoxia. The generated output will not only provide novel insight into the role of ketone bodies under hypoxic conditions but will also be of applied value for mountaineers and athletes competing at altitude as well as for multiple clinical diseases associated with hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 35 years old
* Body Mass Index (BMI) between 18 and 25
* Physically fit and regularly involved in physical activity (2-5 exercise sessions of > 30min per week)
* Good health status confirmed by a medical screening
* Non smoking

Exclusion Criteria:

* Any kind of injury/pathology that is a contra-indication for hypoxic exposure and/or to perform high-intensity exercise
* Intake of any medication or nutritional supplement that is known to affect exercise, performance or sleep
* Intake of analgesics, anti-inflammatory agents, or supplementary antioxidants, from 2 weeks prior to the start of the study.
* Recent residence or training under hypoxia; more than 7 days exposure to altitude > 2000m during a period of 3 months preceding the study.
* Night-shifts or travel across time zones in the month preceding the study
* Blood donation within 3 months prior to the start of the study
* Smoking
* More than 3 alcoholic beverages per day
* Involvement in elite athletic training at a semi-professional or professional level
* Any other argument to believe that the subject is unlikely to successfully complete the full study protocol

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Cerebrovascular reactivity to carbon dioxide (CO2) | On Day 1 at sea level (in normoxia). On Day 2 (36 hours after) of exposure to hypobaric hypoxia.
  Subjects will breathe 4 min 3% CO2 and 4 min 6% CO2 separated by 4 min of breathing ambient air. The middle cerebral artery will be continuously recorded by transcranial Doppler.
Cognitive function | On Day 1 at sea-level (in normoxia). On Day 0 and Day 2 (4 hours and 48 hours) after exposure to hypobaric hypoxia, respectively.
  Cognitive function will be assessed by the computerized psychometric test battery: The Psychology Experiment Building Language (PEBL). The following cognitive tests will be used: The color-stroop test (measures attention, processing speed, and inhibitory control; the time it takes to complete the task and the accuracy of the responses; the number of correct and incorrect responses), the digit-span test (measures an individual's working memory capacity and short-term memory; the score of correctly remembered digit span), the ppvt test (measures the reaction time, attention, concentration; the time to react on the visual signal) the fitts test (measures the hand-eye coordination, fine motor skills, concentration; time to position the target) and the timewall test (measures the reasoning, calculating, reaction time, strategy and problem-solving; estimate the time when a moving target will reach a location behind a wall).
Acute Mountain Sickness (AMS) | Every day at 9.00 p.m. (before sleep) and at 6.15 a.m. (upon waking) in normoxia and hypobaric hypoxia, respectively.
  Acute Mountain Sickness (AMS) will be assessed by the Lake Louise scale. The symptoms measured on the test include headache, gastrointestinal upset, fatigue/weakness, dizziness/light-headedness, and sleep disturbance. These are rated with an intensity level from 0 (the lowest) to 3 (the highest). A total score that is ≥3, including a headache, is indicative of AMS.
Change in lung function estimating forced vital capacity (FVC) and forced expiratory volume in 1st second (FEV1). | On Day 1 at sea level and on Day 3 of exposure to hypobaric hypoxia.
  Lung function will be assessed by FVC and FEV1.
Change in lung function estimating peak expiratory flow (PEF). | On Day 1 at sea level and on Day 3 of exposure to hypobaric hypoxia.
  Lung function will be assessed by PEF.
Change in lung function | On Day 1 at sea level and on Day 3 of exposure to hypobaric hypoxia.
  Lung function will be assessed by the FEV1/FVC ratio.
Heart rate response to exercise | Every day during each 20-90 min long exercise bout performed between 9 a.m. and 6 p.m.. On Day 0 and Day 1 in normoxia. On Day 0, Day 1, Day 2, and Day 3 in hypobaric hypoxia.
  Heart rate (HR, bpm) will be continuously monitored during different exercise bouts of a variety of intensities (moderate and heavy intensities will be used).
Respiratory response to exercise | Every day during each 20-90 min long exercise bout performed between 9 a.m. and 6 p.m.. On Day 0 and Day 1 in normoxia. On Day 0, Day 1, Day 2, and Day 3 in hypobaric hypoxia.
  Oxygen consumption (VO2, L/min and mL/min/kg) will be continuously monitored during different exercise bouts of variety intensities (moderate and heavy intensities will be used).
Changes in muscular oxygenation during exercise | Every day during each 20-90 min long exercise bout performed between 9 a.m. and 6 p.m.. On Day 0 and Day 1 in normoxia. On Day 0, Day 1, Day 2, and Day 3 in hypobaric hypoxia.
  Muscle oxygenation/deoxygenation will be continuously recorded during each exercise bout by Near Infra-Red Spectroscopy (NIRS) placed on the vastus lateralis. NIRS measure the quantity of oxygenated and deoxygenated haemoglobin and myoglobin (microM) in the investigated areas (vastus lateralis).
Changes in cerebral oxygenation during exercise | Every day during each 20-90 min long exercise bout performed between 9 a.m. and 6 p.m.. On Day 0 and Day 1 in normoxia. On Day 0, Day 1, Day 2, and Day 3 in hypobaric hypoxia.
  Brain oxygenation/deoxygenation will be continuously recorded during each exercise bout by Near Infra-Red Spectroscopy (NIRS) placed at the frontal levels. NIRS measure the quantity of oxygenated and deoxygenated haemoglobin (microM) in the investigated areas (prefrontal cortex).
Changes in the rate of muscular oxygen consumption (mV#O2) | Every day before each 20-90 min long exercise bout performed between 9 a.m. and 6 p.m.. On Day 0 and Day 1 in normoxia. On Day 0, Day 1, Day 2, and Day 3 in hypobaric hypoxia.
  Muscle oxygen consumption will be assessed using a previously validated protocol. Briefly, a Near Infra-Red Spectroscopy (NIRS) optode will be placed on the vastus lateralis muscle. Before the protocol, an ischemic calibration will be performed to normalize the NIRS signals by inflating the blood pressure cuff to 250-300 mmHg for a maximum of 5 min. Resting mV#O2 will be assessed from the decrease in muscle oxygenation which accompanies the arterial occlusion.Then, each subject will perform a 3 x 6 minutes moderate-intensity exercise, 8 minutes heavy-intensity exercise and graded exercise test. To measure the recovery of oxygen consumption after exercise, subject will have a series of arterial occlusion as follows: 5 occlusions 5sec on-5sec off, 5 occlusions 5sec on-5sec off, and 5 occlusions 10 sec on-20 sec off.
Duration of different sleep stages | Throughout the entire duration of the night, up to 8 hours after individual bedtime (between 10 p.m. and 6 a.m.). On Day 0 in normoxia. On Day 0 and Day 2 in hypobaric hypoxia.
  Polysomnography will be used to assess the duration of the different sleep stages.
Changes in oxidative stress markers in the blood | Blood samples will be collected on Day 1 in normoxia and Day 1, Day 2 and Day 3 in hypobaric hypoxia at 6 a.m. (upon waking).
  Oxidative stress markers concentration will be measured on collected venous blood sample.
Change in salivary cortisol concentration | Saliva samples will be collected on Day 1 in normoxia and Day 1, Day 2 and Day 3 in hypobaric hypoxia at 6 a.m. (upon waking).
  Cortisol concentration will be measured on collected saliva samples.
Change in hydration status | Urine samples will be collected on Day 1 in normoxia and Day 1, Day 2 and Day 3 in hypobaric hypoxia at 6 a.m. (upon waking).
  Urine samples will be assessed using urine specific gravity.
Baroreflex sensitivity | Within 24 h hours after exposure to normoxia and hypobaric hypoxia, respectively
  At sea level: subjects will breath 6 min normal ambient air (21% O2, 0.03% CO2), 6 hypoxic normocapnic (13.8% O2, 0.03% CO2), and 6 min normoxic hypercapnic (21% O2, 3% CO2) air.
  At high altitude: subjects will breath 6 min hypobaric hypoxic (21% O2, 0.03% CO2), hypobaric normoxic (32% O2, 0.03% CO2), hypobaric normoxic hypercapnic (32% O2, 3% CO2) air.
Change in nocturnal oxygen saturation | Throughout the entire duration of the night, up to 8 hours after individual bedtime (between 10 p.m. and 6 a.m.). On Day 0 in normoxia. On Day 0 and Day 2 in hypobaric hypoxia.
  Measured using pulse oximetry
Absolute amount of nocturnal urinary catecholamine excretion | From 10 p.m. to 6 a.m. on Day 0 in normoxia and Day 0, Day 1 and Day 2 in hypobaric hypoxia.
  Measured using ELISA of collected nocturnal urine. Subjects empty bladder before sleep and urine will be collected throughout the entire duration of the night, up to 8 hours. Up to 8 hours from 10 p.m. to 6 a.m. on Day 0 in normoxia and Day 0, Day 1 and Day 2 in hypobaric hypoxia.

SECONDARY OUTCOMES:
Change in cerebral blood flow in the internal carotid artery | On Day 1 at sea level (in normoxia). On Day 2 (36 hours after) of exposure to hypobaric hypoxia.
  Cerebral blood flow in the internal will be assessed every morning by doppler ultrasound.

CONTACTS AND LOCATIONS:
Locations (2):
- KU Leuven, Leuven, Belgium
- Jozef Stefan Institute, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tominec D, Stalmans M, Narang BJ, Millet GP, Poffe C, Debevec T. Exogenous Ketosis during Early Acclimatization at High Altitude: Ventilatory, Cardiovascular and Muscular Responses to Maximal Exercise. Med Sci Sports Exerc. 2025 Nov 1;57(11):2468-2479. doi: 10.1249/MSS.0000000000003791. Epub 2025 Jun 13. PMID 40523225